CLINICAL TRIAL: NCT01979653
Title: A Comparision of Midazolam-dexmedetomidine With Dexmedetomidine Alone for Hemodynamic Stability and Quality of Sedation in Elderly Patients Under Spinal Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2013-0615
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2013-11

CONDITIONS: Sedation; Aged; Hemodynamics
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine alone (Experimental): dexmedetomidine 0.5 mcg/kg for 10 min + normal saline (volume-matched) bolus + dexmedetomidine 0.2-0.4 mcg/kg/hr infusion
  Interventions: Drug: dexmedetomidine alone or dexmedetomidine + midazolam
- dexmedetomidine + midazolam (Experimental): normal saline (volume-matched) for 10 min + midazolam 0.2 mg/kg bolus + dexmedetomidine 0.2-0.4 mcg/kg/hr infusion
  Interventions: Drug: dexmedetomidine alone or dexmedetomidine + midazolam

INTERVENTIONS:
Drug: dexmedetomidine alone or dexmedetomidine + midazolam

SUMMARY:
The purpose of this study is to compare midazolam-dexmedetomidine with dexmedetomidine alone for hemodynamic stability and quality of sedation in elderly patients under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years
* ASA physical status class I-II
* the patients who want sedation during elective lower limb surgery under spinal anesthesia

Exclusion Criteria:

* contraindication to spinal anesthesia
* neurologic or cognitive dysfunction
* severe cardiovascular or pulmonary disease
* refusal to participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability | 4 hour
  comparison of bradycardia incidence

SECONDARY OUTCOMES:
Modified Observer Assessment of Alertness/Sedation (MOAAS) scale | 4 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea